CLINICAL TRIAL: NCT04298593
Title: Assessment of Arrhythmic BuRdEn With Post-ProCedural COntinuous ElectRocarDiographic Monitoring in Patients Undergoing Transcatheter Aortic Valve Implantation: The RECORD Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Principal Investigator, Josep Rodes-Cabau, MD, Principal investigator, Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RECORD
Record Dates: First submitted 2020-01-12; First posted 2020-03-06 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: TAVI; ECG Monitoring

STUDY DESIGN:
Intervention Model Description: Prospective registry
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ECG monitoring (Other): All patient will be under telemetry
  Interventions: Device: Cardiostat

INTERVENTIONS:
Device: Cardiostat — This is a prospective observational study including patients accepted by the heart team for a TAVI procedure. There will be no restriction regarding the type of valve and approach used for the TAVI procedure. Following the TAVI procedure, the patients will be under telemetry until hospital discharge and, at hospital discharge, they will be monitorized up to 4 more weeks using the CardioSTAT® device.

SUMMARY:
TAVI recipients exhibit a high burden of arrhythmic events early after the procedure. ECG continuous monitoring could be useful to diagnose and facilitate early implementation of specific therapeutic measures in these patients.

DETAILED DESCRIPTION:
Prospective registry including patients accepted by the heart team for a TAVI procedure. Patients will undergo a prolonged continuous ECG monitoring using the CardioSTAT® device after hospital discharge. Following the TAVI procedure, continuous ECG monitoring will start just before hospital discharge and prolonged up to 4 weeks. There won't be any restriction regarding the type of valve and approach used for the TAVI procedure.

All type of arrhythmic events will be recorded, as well as the specific therapeutic measures implemented upon the diagnosis of the arrhythmic event.

Analyses of the CardioSTAT will be done at 2 and 4 weeks following hospital discharge. Clinical follow-up will be performed at 14 days (analysis of CardioSTAT® record), 28 days (analysis of CardioSTAT record), 1 year post-TAVI and yearly thereafter up to 5-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe aortic stenosis undergoing TAVI with either balloon or self-expandable valves.

Exclusion Criteria:

* Failure to provide informed consent.
* Prior or post-procedural pacemaker
* In-hospital death
* Logistic reasons precluding ECG monitoring within the 4 weeks after the procedure
* Participation in another continuous ECG monitoring post-TAVI trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-06-28 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of arrhythmic events | within the first weeks after the procedure, an average of 4 weeks
  Incidence of arrhythmic events after discharge in TAVI recipients.
Type of arrhythmic events | within the first weeks after the procedure, an average of 4 weeks
  Type of arrhythmic events after discharge in TAVI recipients.
Incidence of arrhythmic events and treatment modification | within the first weeks after the procedure, an average of 4 weeks
  Incidence of arrhythmic events leading to a specific change in treatment.
Type of arrhythmic events and treatment modification | within the first weeks after the procedure, an average of 4 weeks
  Type of arrhythmic events leading to a specific change in treatment.

SECONDARY OUTCOMES:
Number of participants with pacemaker | Through study completion, an average of 5 years
  Incidence of permanent pacemaker implantation after the procedure.
Number of participants with treatment modification | Through study completion, an average of 5 years
  Number of participants who required change in their medication (anticoagulation, antiarrhythmic) after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- IUCPQ, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baumgartner H, Falk V, Bax JJ, De Bonis M, Hamm C, Holm PJ, Iung B, Lancellotti P, Lansac E, Munoz DR, Rosenhek R, Sjogren J, Mas PT, Vahanian A, Walther T, Wendler O, Windecker S, Zamorano JL. 2017 ESC/EACTS Guidelines for the Management of Valvular Heart Disease. Rev Esp Cardiol (Engl Ed). 2018 Feb;71(2):110. doi: 10.1016/j.rec.2017.12.013. No abstract available. English, Spanish. PMID 29425605
- [Background] Auffret V, Puri R, Urena M, Chamandi C, Rodriguez-Gabella T, Philippon F, Rodes-Cabau J. Conduction Disturbances After Transcatheter Aortic Valve Replacement: Current Status and Future Perspectives. Circulation. 2017 Sep 12;136(11):1049-1069. doi: 10.1161/CIRCULATIONAHA.117.028352. PMID 28893961
- [Background] Urena M, Rodes-Cabau J. Conduction Abnormalities: The True Achilles' Heel of Transcatheter Aortic Valve Replacement? JACC Cardiovasc Interv. 2016 Nov 14;9(21):2217-2219. doi: 10.1016/j.jcin.2016.09.040. No abstract available. PMID 27832847
- [Background] Moreno R, Dobarro D, Lopez de Sa E, Prieto M, Morales C, Calvo Orbe L, Moreno-Gomez I, Filgueiras D, Sanchez-Recalde A, Galeote G, Jimenez-Valero S, Lopez-Sendon JL. Cause of complete atrioventricular block after percutaneous aortic valve implantation: insights from a necropsy study. Circulation. 2009 Aug 4;120(5):e29-30. doi: 10.1161/CIRCULATIONAHA.109.849281. No abstract available. PMID 19652115
- [Background] Siontis GCM, Praz F, Lanz J, Vollenbroich R, Roten L, Stortecky S, Raber L, Windecker S, Pilgrim T. New-onset arrhythmias following transcatheter aortic valve implantation: a systematic review and meta-analysis. Heart. 2018 Jul;104(14):1208-1215. doi: 10.1136/heartjnl-2017-312310. Epub 2017 Dec 23. PMID 29275399
- [Background] Rodes-Cabau J, Urena M, Nombela-Franco L, Amat-Santos I, Kleiman N, Munoz-Garcia A, Atienza F, Serra V, Deyell MW, Veiga-Fernandez G, Masson JB, Canadas-Godoy V, Himbert D, Castrodeza J, Elizaga J, Francisco Pascual J, Webb JG, de la Torre JM, Asmarats L, Pelletier-Beaumont E, Philippon F. Arrhythmic Burden as Determined by Ambulatory Continuous Cardiac Monitoring in Patients With New-Onset Persistent Left Bundle Branch Block Following Transcatheter Aortic Valve Replacement: The MARE Study. JACC Cardiovasc Interv. 2018 Aug 13;11(15):1495-1505. doi: 10.1016/j.jcin.2018.04.016. Epub 2018 Jul 18. PMID 30031719
- [Background] Mautner RK, Phillips JH. Atrioventricular and intraventricular conduction disturbances in aortic valvular disease. South Med J. 1980 May;73(5):572-8, 581. doi: 10.1097/00007611-198005000-00008. PMID 7375971
- [Background] Widgren V, Dencker M, Juhlin T, Platonov P, Willenheimer R. Aortic stenosis and mitral regurgitation as predictors of atrial fibrillation during 11 years of follow-up. BMC Cardiovasc Disord. 2012 Oct 18;12:92. doi: 10.1186/1471-2261-12-92. PMID 23075140
- [Background] MacMillan RM, Demorizi NM, Gessman LJ, Maranhao V. Correlates of prolonged HV conduction in aortic stenosis. Am Heart J. 1985 Jul;110(1 Pt 1):56-60. doi: 10.1016/0002-8703(85)90514-9. PMID 4013990